CLINICAL TRIAL: NCT04463446
Title: The Impact of an Innovative eHealth Transition Intervention on Self-Management Skills Among Young Adults With Congenital Heart Disease
Acronym: READYorNot CHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: McGill University (Other); Oregon Health and Science University (Other); University of British Columbia (Other); University of Toronto (Other); Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00097233
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Congenital Heart Disease; Congenital Heart Disease in Adolescence
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The app arm (Experimental): Use of CHD app
  Interventions: Behavioral: Use of the CHD app
- Nurse-led intervention arm (Active Comparator): Nurse-led intervention
  Interventions: Behavioral: Nurse-led intervention

INTERVENTIONS:
Behavioral: Use of the CHD app — Use of the CHD app
  Arms: The app arm
Behavioral: Nurse-led intervention — Teaching session with clinic nurse
  Arms: Nurse-led intervention arm

SUMMARY:
Congenital heart disease (CHD) survivors constitute one of the fastest growing populations in adult cardiology practices. This population is vulnerable to gaps in care, particularly as they graduate from the pediatric to adult healthcare system. Their healthcare needs are complex, and preparing this population for transfer to adult care is a resource-intense process.

This trial will evaluate the use of the MyREADY Transition CHD app against a nurse-led one-time intervention in clinic. Participants will be 16-17 year olds who attend a cardiology outpatient clinic. The app will allow young adults to learn about their heart condition and about self-management skills in the context of adult healthcare by using the app for 18 months. The nurse-led intervention will cover similar topics, but in a one-time in-person session with a clinic nurse.

Outcomes: The primary outcome is change in Transition Readiness Assessment Questionnaire (TRAQ) score over time. Secondary outcomes are change in the MyHeart Score and the General Self-Efficacy (GSE) score. These questionnaires will be answered by all participants at regular intervals (enrollment, 1 month, 6 months, 12 months, 18 months) throughout the trial. The trial will also consider time to the first adult cardiology appointment, cost of the interventions, and will conduct interviews with participants in the app group to learn about their experiences using the app.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) survivors constitute one of the fastest growing populations in adult cardiology practices. This population is vulnerable to gaps in care, particularly as they graduate from the pediatric to adult healthcare system, yet their healthcare needs are complex, costly, and chronic. With this submission, we focus on transitions in care (TiC) from pediatric to adult healthcare with a research plan designed to optimize TiC outcomes. Despite universal health insurance, clinical programs have insufficient resources to provide transition preparation for adolescents with cardiac disease. This likely reflects a lack of human and financial resources, geographic distance for patients and families living in rural communities, and/or a "process" problem wherein no one is directly accountable for transition. Nonetheless, Canadian policy mandates transfer to the adult healthcare system at age 18 regardless of transition readiness.

2.1 Design. Cluster RCT with 2 arms conducted in accordance with CONSORT guidelines within a mixed methods convergent design. The cluster design will minimize cross-contamination. The qualitative and quantitative data will be collected concurrently, and the data merged to ensure that intervention effectiveness is fully understood.

2.2 Planned trial interventions. This study will compare (i) access to the app vs. our team's established 1-on-1 nurse-led TiC intervention.

The App: Content of the app will be developed during Phase 1 in conjunction with the PFAC. A study registered nurse (RN) will orient participants to the app, provide them with a unique username and password, and help them create an individualized MyHealth passport (note that CHD transition guidelines recommend the use of health passports). The anticipated duration is 30 minutes. A research assistant (RA) will be available to participants throughout the study period to answer questions about the app. System-generated automatic text messages will be sent to participants every month to remind them about the app. The RA will check in with participants every 3 months. Those who do not use the app over a 3-month period will be flagged to identify psychological and environmental barriers to app use.

Nurse-led TiC intervention: There will be two cardiology RNs, each with adolescent experience, at each site who are different from the RN working with participants in the app group, to avoid cross contamination. The intervention will be provided during a single 60-75 minute session with the RN; this was the time required in the CHAPTER 1 and 2 Studies. Sessions will occur on the same day as a clinic appointment. Sessions will be interactive and engaging. Individual sessions, in contrast to a group, allow for the content to be participant-specific and at a pace compatible with the participant and their cognitive and social abilities. This intervention, already refined by our study team, will focus on increasing knowledge about the adolescent's CHD and promotion of self-management and self-efficacy skills.

Prior to the session, the RN will review the medical record to become familiar with the participant's cardiac history. The intervention addresses both education about the participant's CHD (steps i-v) and self-management skills (steps vi-viii). Specific elements include: (i) introduction to transition and its importance, (ii) creation of a MyHealth Passport, including name of CHD, prior cardiac interventions, and healthcare provider contact information, (iii) diagram of participant's cardiac anatomy, (iv) discussion of three potential future cardiac complications that are diagnosis-specific and individualized, (v) introduction to the iHeartChange CHD transition website (iheartchange.org) developed by team member Kovacs, (vi) discussion of the concept of self-management, (vii) viewing and discussion of three professionally developed 1-minute videos that demonstrate interactions between a healthcare provider and a young adult with poor communication skills (i.e., what went wrong, how to handle this better) and three 1-minute videos demonstrating assertive communication skills (i.e., strengths, successes), and (viii) adolescent practice of a "3-sentence summary" about their CHD, with feedback from the RN.

Nurse-led intervention fidelity and quality assurance (Nurse-led intervention group only). This will be performed in the same manner as the CHAPTER 2 study. Months 13-15 will be a quality assurance (QA) phase. Role-modeling of an intervention with a standardized patient will be led by team member Kovacs, who will provide in-person training to study RNs. Each RN will then practice with a standardized patient with audio taping for review and feedback by Kovacs and Dimitropoulos. Subsequently, 20 participants will be enrolled and receive the intervention (2 patients per study RN x 2 RNs per site x 5 study sites). These sessions will also be audio taped with participant permission. After each session the RN will complete a fidelity checklist and nursing intervention log to record completion of each intervention component as described above. Nurse-generated field notes will record RN's observations of their interactions with adolescents, including the adolescent's confidence, engagement, and emotional responses. Sessions will be digitally audio-recorded with participant permission; 1/5 will be randomly selected for evaluation of treatment fidelity. Evaluation of treatment fidelity will be based on review of nursing intervention logs, fidelity checklists, field notes and audiotapes monthly by Kovacs and Dimitropoulos. Participants enrolled from months 16-27 inclusive will contribute to study outcomes.

2.3 Group allocation. Participants will be randomized by clusters defined by week of attendance in the pediatric cardiology clinic, as per CHAPTER 1 and 2 Studies. As week (rather than individual participant) is the unit of randomization, this is a cluster randomization design. This method of randomization prevents two adolescents in the same waiting room being allocated to different groups, with adolescents in the app group potentially preferring to be in the nurse intervention group (or vice-versa). Each cardiologist has a weekly clinic and therefore a given cardiologist's patients will be allocated to each study arm equally, preventing potential bias by cardiologist co-intervention. We anticipate average enrolment of 1-2 participants per site per week, i.e. cluster size will be ≤ 2. To determine "app weeks" vs. "nurse intervention weeks", a biostatistician will prepare the randomization sequence. Permuted-block randomization with varying block sizes and equal allocation ratio will be used to ensure balanced allocation of weeks (randomization unit) between the 2 treatment arms. Blocks of sizes 2 and 4 will be randomly mixed to overcome the problem of predicting the allocation for the last few entries in each block. Since five centers are participating in the trial, a randomization schedule will be provided for each center.Randomization will be stratified by center to ensure a similar number of participants are allocated to each group within each site; this will mitigate the potential impact of center-specific confounders.

2.4 Protecting against sources of bias. Participants, their parents, and study RNs will be aware of group allocation as blinding is not feasible. However, adolescents and parents in both groups will be unaware of the primary outcome and therefore will not be able to consciously influence this outcome. Intervention occurs on the same day as a clinic appointment, but clinic RNs and pediatric cardiologists will not be informed of group allocation, and this approach has been feasible in the CHAPTER 1 and CHAPTER 2 studies. Study RNs will be instructed to not inform clinicians of app vs. nurse-intervention weeks.

2.5 Inclusion/exclusion criteria: described elsewhere

2.6 Duration of intervention. As per section 2.2, participants in the app group will meet with an RN for ~30 min and then have access to the app for ~ 18 months. Participants in the nursing intervention will meet once with a study RN (60±15 min). All RN contact will be coordinated with a clinic appointment.

2.7 Frequency and duration of follow-up. Participants in both groups will complete questionnaires at enrollment (baseline), 1, 6, 12, and 18 months post enrollment (see below). Eighteen months was chosen because our CHAPTER 1 and 2 studies yielded benefits at or before this time.

2.9 Measurement of outcomes at follow-up. Participants will complete follow-up online questionnaires at home, independently of their parents. For adolescents not having home Internet access, we will arrange for access via their school or local library. Adolescents not completing the follow-up questionnaires will be contacted by mail, email, or text (depending on their preference) every 2 weeks for a total of 3 times, and then telephoned once, to be reminded. A $25 gift card (iTunes, Tim Hortons or Amazon) will be provided to participants at each time point to acknowledge their time and commitment to questionnaire completion.

ELIGIBILITY:
Inclusion Criteria:

* moderate or complex CHD
* seen at outpatient cardiology clinic at participating pediatric hospital

Exclusion Criteria:

* < Grade 6 level of reading and comprehension
* heart transplantation

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Transition Readiness Assessment Questionnaire | 18 months
  The Transition Readiness Assessment Questionnaire contains a series of questions in which the youth is asked to describe their ability level in various skill areas related to their health and health care, using the following scale:
  No, I do not know how No, but I want to learn No, but I am learning to do this Yes, I have started doing this Yes, I always do this when I need to
  This produces a minimum score 20, max score 100. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
MyHeart Score | 18 months
  The MyHeart Scale assess CHD knowledge. Score is 0-100, a higher score indicates a better outcome.
General Self-Efficacy Score | 18 months
  The scale was created to assess a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events. Score is between 10-40, a higher score insicates a better outcome.

OTHER OUTCOMES:
Excess time to adult care | 18 months
  The recommended time to first adult cardiology appointment will be compared to the actual time to first adult cardiology appointment. Participants who have not attended the adult clinic by the end of the study period (i.e., are "censored") will still contribute to this outcome as survival analysis is designed to accommodate censored data. Delays in attending the adult clinic related to system factors (e.g. waiting list) will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mackie, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada